CLINICAL TRIAL: NCT05267899
Title: A Phase I, First in Human, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of WGI-0301, a Lipid Nanoparticle Suspension of Akt-1 Antisense Oligonucleotide, in Patients With Advanced Solid Tumors
Brief Title: A Phase I First in Human Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of WGI-0301 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Haichang Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WGI0301-P1U
Record Dates: First submitted 2022-02-08; First posted 2022-03-07 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- WGI-0301 (Experimental)
  Interventions: Drug: WGI-0301

INTERVENTIONS:
Drug: WGI-0301 — WGI-0301 is a lipid nanoparticle preparation of Archexin® for the treatment of advanced solid tumors.

SUMMARY:
The purpose of this study is to learn about the effects of a study medicine, WGI-0301 to find the best dose for treating solid tumors, and to see how safe and tolerable the study drug is for patients with solid tumors.

The study is also done to learn how the study drug is taken up by your body; this is called Pharmacokinetic (PK) studies and how the study drug affects the body; this is called Pharmacodynamics (PD)

ELIGIBILITY:
Inclusion Criteria Subjects must meet all the following criteria to participate this study

1. Subject with measurable disease based on RECIST 1.1.
2. Advanced, histologically or cytologically confirmed solid tumors who have progressed from current therapy or who have relapsed after prior therapy and are not candidates for potentially curative therapy.
3. Pathologically confirmed solid tumors.
4. Patients with advanced solid tumors (unresectable or metastatic) who failed standard therapy (disease progression or intolerance).
5. Capable of understanding the written informed consent, provides signed, dated, and witnessed written informed consent, and agrees to comply with the study protocol.
6. Age 18 years or older at first screening/ examination visit.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2, measured within 72 hours of 1st treatment.
8. Adequate hematological function [absolute neutrophil count (ANC) ≥ 1.5 × 109/L], [Platelets ≥ 100 × 109/L], [Hemoglobin ≥ 9 g/dL], and [Serum albumin ≥ 2.8 g/dL].
9. Adequate renal function [calculated estimate glomerular filtration rate (eGFR) of ≥ 50mL/min] using the CKD-EPI Creatinine Equation (2021).
10. Adequate hepatic function [total bilirubin ≤ 1.5 x UNL; AST (aspartate transaminase) or ALT (alanine transaminase) ≤ 3 x UNL or ≤ 5 x UNL if due to liver involvement by tumor.
11. Negative pregnancy test for women of child-bearing potential (WOCBP) and males need to agree to use a highly effective method of contraception if not surgically sterile prior to study entry, while on drug, and for 3 months' time after the last dose. Please refer to Appendix 1 for acceptable effective contraceptive methods.
12. Subject who has predicted life expectancy of at least 12 weeks.

Exclusion Criteria Subjects meet one or more of below criteria will be excluded

1. Lactating, pregnant, or intend to be pregnant.
2. Received anti-cancer therapy or other investigational drugs within 4 weeks prior to the 1st dose of study drug.
3. Patient in use of sensitive substrates of major cytochrome P450 enzymes and transporters based on FDA Drug Development and Drug Interactions, Table of Substrates, Inhibitors, and Inducers, or strong inducers of transporter, P-gp, including apalutamide, carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, St. John's wort. Patient in use of strong inhibitors of transporters based on based on FDA Drug Development and Drug Interactions, Table of Substrates, Inhibitors, and Inducers (Appendix 2).
4. All acute toxic effect of any prior antitumor therapy resolved to Grade 1 before the start of study therapy (with the exception of alopecia [G 1 or 2 permitted], neurotoxicity [Grade ≤ 2 permitted], or selected lab parameters [Grade < 2 permitted with exceptions noted below].
5. Has evidence of another malignancy not in remission or history of such a malignancy within the last 3 years (except for treated basal or squamous cell carcinoma of the skin, or in situ cancer of the cervix). Concomitant malignancies except carcinoma in situ, basal or squamous cell skin carcinoma; low grade prostate cancer treated with prostatectomy more than 5 years ago; early-stage melanoma treated with complete surgical excision more than 5 years ago; carcinoma in situ of cervix treated with cone procedure more than 8 years ago.
6. Has symptomatic central nervous system (CNS) metastases, except where metastases are stable over a three-month period.
7. Has unstable bleeding disorder or currently under non-established course of anticoagulant therapy (except for the use of heparinized saline to maintain the patency of central venous catheters).
8. Has a medical history of symptomatic CHF (New York Heart Association [NYHA] classes II-IV) or serious cardiac arrhythmia requiring treatment.
9. Has a medical history of myocardial infarction or unstable angina within 6 months before registration.
10. Has a QTcF prolongation to > 470 ms based on a 12-lead ECG in triplicate, or other abnormalities that in the opinion of the Investigator increase the risk of participating in the study.
11. Has higher or equal to Grade 3 hypertension (≥ 160/100 mmHg) or ≤ 80/50 mmHg; has heart rate (HR) ≥ 100 beats per minute (bpm), or ≤ 45 bpm, confirmed by a repeat assessment.
12. Has evidence of electrolyte imbalance such as hypokalemia, hypocalcemia, and hypomagnesaemia of NCI-CTCAE Grade ≥ 2 (symptomatic, intervention indicated).
13. Major surgery besides tumor resection, within 4 weeks prior to screening
14. Has uncontrolled diabetes mellitus, neurologic or psychiatric condition, an ongoing systemic (including opportunistic) clinically significant infections or any other significant or unstable concurrent medical illness that may increase the risk of study participants determined by Investigator.
15. Has a known history of human immunodeficiency virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Approximately 16 months
  Incidence and severity of treatment-related adverse events and serious adverse events
Recommended Phase 2 Dose of WGI-0301 | Approximately 16 months
  Based on dose-limiting toxicities, the maximal tolerated dose and all other available safety, pharmacokinetic/pharmacodynamic data as assessed by the cohort review committee

SECONDARY OUTCOMES:
Area under the curve | Approximately 16 months
  Area under the plasma concentration time curve of WGI-0301
Maximum plasma concentration | Approximately 16 months
  Highest observed plasma concentration of WGI-0301
Time of maximum plasma concentration | Approximately 16 months
  Time to reach highest observed plasma concentration of WGI-0301
Half-life | Approximately 16 months
  Plasma concentration half-life of WGI-0301

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Valkyrie Clinical Trials, Los Angeles, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No